CLINICAL TRIAL: NCT06159595
Title: Behavioral and Neuronal Correlates of Human Mood States
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Corey Keller, Principal Investigator, Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 11354-2; 1R21MH134172 (NIH)
Record Dates: First submitted 2023-11-16; First posted 2023-12-07 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder; Epilepsy
MeSH Terms: conditions — Depressive Disorder, Major; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Direct electrical stimulation (DES) (Active Comparator): Intracranial electrodes will be used for the delivery of invasive brain stimulation.
  Interventions: Device: Intracranial electrodes
- Sham Direct electrical stimulation (DES) (Sham Comparator): Intracranial electrodes will be used for the delivery of invasive brain stimulation.
  Interventions: Device: Intracranial electrodes

INTERVENTIONS:
Device: Intracranial electrodes — Surgically-implanted intracranial electrodes.

SUMMARY:
Optimizing treatments in mental health requires an easy to obtain, continuous, and objective measure of internal mood. Unfortunately, current standard-of-care clinical scales are sparsely sampled, subject to recency bias, underutilized, and are not validated for acute mood monitoring. The recent shift to remote care also requires novel methods to measure internal mood. Recent advances in computer vision have allowed the accurate quantification of observable speech patterns and facial representations. The continuous and objective nature of these audio-facial behavioral outputs also enable the study of their neural correlates. Here, the investigators hypothesize that video-derived audio-facial behaviors have discrete neural representations in the limbic network and can provide a critical set of reliable longitudinal estimates of mood at low cost across home and clinic settings.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 and 65
* Major depressive disorder (MDD) in a current major depressive episode diagnosed with the Mini-International Neuropsychiatric Interview (MINI)
* No medical or surgical contraindication to electrode implantation
* Patient capable of understanding the scope of our project or signing informed consent independently.

Exclusion Criteria:

* Diffuse epilepsy involving several lobes of the brain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Quantitative Audio-Facial Change | 5 minutes
  Quantitative percent change in each audio-facial feature before and after direct electrical stimulation at each site.
Quantitative Mood Change | 5 minutes
  Quantitative percent change in Immediate Mood Scaler (IMS) after direct electrical stimulation at each site compared to a baseline period before sham. The minimum score on the IMS is 7 and the maximum is 154, with lower scores reflecting more negative mood states.

SECONDARY OUTCOMES:
Correlation between Audio-Facial and Mood Change | 5 minutes
  Quantitative audio facial changes will be compared to quantitative changes in mood at each site by means of correlation and binary comparisons.
Qualitative Mood Change | 5 minutes
  Qualitative articulation of mood (participants freely articulate mood after direct electrical stimulation at each site) and speech transcripts will be analyzed for ratio of positive and negative valence words.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States